CLINICAL TRIAL: NCT05241990
Title: A Hybrid Type III Implementation Trial Testing Practice Facilitation as a Strategy to Improve Alcohol Treatment Adoption and Implementation in HIV Care
Brief Title: Practice Facilitation as a Strategy to Improve Alcohol Treatment Adoption and Implementation in HIV Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Washington (Other); University of Alabama at Birmingham (Other); Fenway Community Health (Other); University of North Carolina (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00303116; P01AA029544 (NIH)
Record Dates: First submitted 2022-02-07; First posted 2022-02-16 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Hiv; Alcohol Use, Unspecified
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol Drinking | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol Stepped Care (Experimental): Based on severity of alcohol use, individuals receive brief alcohol intervention delivered in person or by computer, cognitive behavioral therapy by person or computer, or pharmacotherapy for alcohol use disorder
  Interventions: Behavioral: Practice Facilitation; Behavioral: Alcohol Stepped Care

INTERVENTIONS:
Behavioral: Practice Facilitation — A practice coach will offer tools, resources, hands-on guidance, and content expertise to assist sites in offering a stepped care model of alcohol treatment to patients with unhealthy alcohol use.
Behavioral: Alcohol Stepped Care — Based on severity of alcohol use, individuals receive brief alcohol intervention delivered in person or by computer, cognitive behavioral therapy by person or computer, or pharmacotherapy for alcohol use disorder

SUMMARY:
Despite availability of evidence-based alcohol reduction interventions (EBI), unhealthy alcohol use remains a barrier to HIV medication adherence, viral suppression and retention in HIV care and consequently HIV treatment as prevention (TASP). Guided by complementary implementation and evaluation frameworks-the Consolidated Framework for Implementation Research (CFIR) and RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance), The investigators will conduct a Hybrid Type 3 effectiveness-implementation evaluating implementation trial testing whether practice facilitation, an evidence-based multifaceted implementation strategy increases reach, adoption, implementation, and maintenance of stepped care for unhealthy alcohol use in three Center for AIDS Research (CFAR) Network of Integrated Clinical Systems (CNICS) HIV clinics located in Boston, San Diego, and Chapel Hill. The investigators will secondarily test whether practice facilitation is associated with decreased unhealthy alcohol use, and improved Antiretroviral Therapy (ART) adherence and viral suppression at the patient level. In practice facilitation, a practice coach will offer tools, resources, hands-on guidance, and content expertise to assist sites in offering a stepped care model of alcohol treatment to patients with unhealthy alcohol use. Stepped care will include brief intervention, cognitive behavioral therapy, and alcohol pharmacotherapy. The practice facilitation intervention will be rolled out sequentially across sites. There will be three phases at each site: pre-implementation planning, implementation with formative evaluation, and post-implementation summative evaluation. Using mixed methods, The investigators specifically propose to meet the following specific aims: (Aim 1) Tailor the practice facilitation intervention to each site using mixed methods (pre-implementation); (Aim 2a) Determine the effects of practice facilitation on implementation of stepped care (primary) and alcohol use and HIV-related outcomes (secondary) using interrupted time series analysis with synthetic controls (summative evaluation); (Aim 2b) Determine the effect of practice facilitation on reach, adoption, and maintenance of evidence-based alcohol treatment using mixed methods (formative evaluation); and (Aim 3) Describe barriers and facilitators to implementation of alcohol-related interventions at each site to describe maintenance and inform widespread sustainable implementation.

ELIGIBILITY:
Inclusion Criteria: Clinic Staff

* Age > 18 years old
* Confirmed to be clinic staff (clinical or administrative roles).
* English speaking
* Cognitively able to complete required survey or interview activities.

Exclusion Criteria Clinic Staff

* Unable to speak English

Inclusion Criteria, Patients

* Confirmed to be a person with HIV (PWH) receiving HIV care and participating in CNICS at one of the three clinic sites
* Scoring AUDIT-C ≥3 for women or ≥4 for men, transgender women or men indicating unhealthy alcohol use.
* Age ≥ 18 years old.
* English speaking.
* Cognitively able to participate in stepped care for unhealthy alcohol use.

Exclusion Criteria, Patients

* Scoring AUDIT-C <3 for women or <4 for men or <4 for transgender women or men
* Age < 18 years old
* Participants cognitively unable to participate in the stepped care for unhealthy alcohol use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Implementation as assessed by the percent of patients receiving an alcohol intervention | 12 months
  Percent of patients receiving an alcohol intervention since their last visit among all eligible individuals.

SECONDARY OUTCOMES:
Change in unhealthy alcohol use as assessed by the Alcohol Use Disorder Identification test-Consumption (AUDIT-C) | Baseline and 12 months
  AUDIT-C Score of <3 in women and <4 in men indicating reduction to lower risk use
Antiretroviral therapy adherence as assessed by a self report on a visual analog scale | 12 months
  Self report of >90% adherence on visual analog scale with higher scores indicating greater adherence
Viral Suppression as assessed by HIV-RNA copies | 12 months
  Viral Suppression will assessed by HIV-RNA copies. HIV-RNA <200 copies indicates viral suppression.

CONTACTS AND LOCATIONS:
Overall Officials: Geetanjali Chander, MD, Principal Investigator — Johns Hopkins University; Betsy McCaul, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- United States (3):
  - University of California, San Diego, San Diego, California
  - Fenway Community Health, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Per NIAAA policy, data will be deposited in the NIAAA Data Archive (NIAAADA), a data repository in the National Institute of Mental Health (NIMH) Data Archive (NDA)
Time Frame: 12 months after study completion
Access Criteria: https://nda.nih.gov/niaaa
URL: https://nda.nih.gov/niaaa